CLINICAL TRIAL: NCT01824641
Title: The Randomized Physiologic Assessment of Thrombus Aspiration in Patients With Acute ST-segment Elevation Myocardial Infarction Trial
Brief Title: Physiologic Assessment of Thrombus Aspiration in Acute ST-segment Elevation Myocardial Infarction Patients
Acronym: PATA-STEMI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: Center of nuclear medicine (Unknown); Institute for histology (Unknown)
Responsible Party: Principal Investigator, Dejan Orlic, MD, Clinical Centre of Serbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T113E4
Record Dates: First submitted 2013-03-22; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Myocardial Infarction
Keywords: Acute myocardial infarction; Manual thrombus aspiration; Coronary physiology
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eliminate (Experimental): Eliminate aspiration catheter
  Interventions: Device: Eliminate aspiration catheter
- Conventional primary angioplasty (Active Comparator): Patients treated with conventional primary angioplasty
  Interventions: Procedure: Conventional primary angioplasty

INTERVENTIONS:
Device: Eliminate aspiration catheter — Eliminate aspiration catheter
  Arms: Eliminate
Procedure: Conventional primary angioplasty — Primary angioplasty without thrombus aspiration
  Arms: Conventional primary angioplasty

SUMMARY:
The Physiologic Assessment of Thrombus Aspiration in ST-segment Elevation Myocardial Infarction (PATA-STEMI) trial is a single center, prospective, randomized trial with a planned inclusion of 128 patients with the first ST-segment elevation myocardial infarction (STEMI). Patients are, before coronary angiography, randomly assigned to thrombus aspiration using 6 or 7 French Eliminate aspiration catheter (Terumo Medical Supply, Japan) or to conventional primary percutaneous coronary intervention (PCI). The primary endpoint is index of microcirculatory resistance (IMR), measured in infarct-related artery, in thrombus aspiration compared to conventional PCI group.

DETAILED DESCRIPTION:
Background and Objective Routine thrombus aspiration is superior to conventional primary PCI in terms of improved myocardial perfusion in STEMI patients. However, myocardial perfusion after thrombus aspiration has not been evaluated by a quantitative, invasive method. Investigators intend to determine whether thrombus aspiration of the infarct-related artery increases myocardial perfusion, as measured by IMR, compared to conventional primary PCI.

Study design PATA-STEMI is a single center, prospective, randomized trial with a planned inclusion of 128 patients with the first STEMI. Patients are randomly assigned, before coronary angiography, to thrombus aspiration using the 6 or 7 French Eliminate aspiration catheter (Terumo Medical Supply, Japan) or to conventional primary PCI. The IMR will be determined in infarct-related artery and non-infarct-related arteries without critical stenosis to measure microcirculatory resistance. The primary endpoint is defined as IMR in infarct-related artery in thrombus aspiration compared to conventional PCI group. Secondary end points are myocardial perfusion grade and resolution of ST-segment elevation, infarct size and left ventricle remodeling, as assessed by echocardiographic indices. Transthoracic echocardiography will be conducted within 24 hours and at 4 months after the primary PCI.

Implications: If manual thrombus aspiration reduces microcirculatory resistance, indicating improved myocardial perfusion, as compared to conventional PCI, it might become the preferred strategy in patients with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with STEMI
* chest pain onset ≤12h, or >12 h with persistent ST-segment elevation
* hemodynamically stable patients

Exclusion Criteria:

* patients without diagnosis of STEMI (pericarditis, for example)
* no written informed consent obtained
* prior Q or non-Q MI
* prior resuscitation
* prior thrombolysis
* prior surgical myocardial revascularisation
* life expectancy <6 months
* periprocedural death

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-05 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
IMR (mmHg seconds) in thrombus aspiration compared to conventional PCI group | At the end of the primary PCI , an expected average of 45 minutes after sheath insertion
  IMR will be measured after final balloon inflation or stent implantation, an expected average of 45 minutes after sheath insertion

SECONDARY OUTCOMES:
Resolution of ST-segment elevation | at 60 minutes after guiding catheter removal
  ST-segment resolution ≥70% at 60 minutes after guiding catheter removal
myocardial blush grade (0-3) | at final angiogram, an expected average of 55 minutes after sheath insertion
  myocardial blush grade will be assessed after IMR measurements, following the final balloon inflation or stent implantation, an expected average of 55 minutes after sheath insertion
infarct size assessed by peak enzyme release (Troponin, creatine kinase MB (CK-MB)) | in hospital course after primary PCI, an expected average of 5 days
  infarct size will be determined based on peak enzyme release (Troponin, CK-MB) during in-hospital stay, an expected average of 5 days
indices of left ventricle remodeling on Echocardiography | within 24 hours and at 4 months after primary PCI
  left ventricle remodeling will be assessed on Echocardiography within 24 hours and at 4 months after primary PCI
infarct size determined by SPECT | within 7-14 days and at 4 months after primary PCI
  infarct size will be determined by SPECT within 7-14 days and at 4 months after primary PCI

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Orlic, MD, Principal Investigator — Clinical Center of Serbia
Locations (2):
- Serbia (2):
  - Clinical center of Serbia, Belgrade
  - Clinical Center of Serbia, Belgrade